CLINICAL TRIAL: NCT00447551
Title: Canadian Study of the Use of Injectable POLY-L-LACTIC Acid (Sculptra Therapy) in Aesthetic Medicine
Brief Title: Canadian Aesthetic Experience With Sculptra Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POLYL_L_01777
Record Dates: First submitted 2007-03-13; First posted 2007-03-14 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Skin Aging
Keywords: Aesthetic facial volume enhancement
MeSH Terms: interventions — poly(lactide); New-Fill

ARMS (1):
- single group (Experimental)
  Interventions: Drug: Poly-L-Lactic Acid

INTERVENTIONS:
Drug: Poly-L-Lactic Acid — Deep dermal injection
  Other Names: Sculptra

SUMMARY:
Primary objective To evaluate the degree of correction achievable with Sculptra for nasolabial folds, mid- and lower facial volume loss, jawline laxity and other signs of facial ageing.

To document the types and incidence of device-related adverse events with Sculptra.

ELIGIBILITY:
Inclusion Criteria:

* Present with nasolabial folds, mid- and lower facial volume loss, jawline laxity or other signs of facial ageing to be treated with Sculptra
* The subject must be willing and able to provide written informed consent that includes a release for use of their photographs in publications. Subjects who refuse the photo release will not be eligible to participate in the study.
* Female subjects must be post-menopausal for at least one year or have had a hysterectomy or tubal ligation; if of child-bearing potential, must agree to use an approved method of birth control throughout the study (i.e., oral/systemic contraceptives, intrauterine device (IUD), or spermicide in combination with a barrier method of contraception);

Exclusion Criteria:

* Personal history of allergic/anaphylactic reactions, including hypersensitivity to local anaesthetics (lidocaine);
* Known history of bleeding disorders;
* Active inflammatory process in the area to be treated (skin eruptions such as cysts, pimples, rashes, cancerous/pre-cancerous lesions, or any other active skin disease);
* Active hepatitis within the past year;
* Subjects who are pregnant or who plan to become pregnant within the study timeframe, or who are breastfeeding;
* HIV positive patients;
* Recent history of trauma in the face (< 1 year);
* Previous use of Dermalive or Dermadeep;
* Previous facial surgery within the last six months;
* Recent facial filler within the last six months;
* Planned surgical interventions (such as rhinoplasty, facelift, congenital defect repair) or use of other fillers or lasers for the initial six months post-Sculptra therapy;
* Subjects with clinically important disease as judged by the investigator within 3 months of the start of the study (e.g., history of significant lab abnormalities, myocardial infarct, stroke, cancer, connective tissue disease, etc.), including subjects with medical conditions that might require the use of immunosuppressive medications during the trial (severe asthma, rheumatoid arthritis, organ transplant, etc.);
* Subjects who have used superficial dermal resurfacing procedures in the facial area, including chemical peel, dermabrasion, or microderm treatments within six weeks of visit 1 and for the duration of the main study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2007-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the degree of correction attainable with Sculptra (injectable PLLA) for the correction of nasolabial folds, mid-and lower facial volume loss, jawline laxicity, and other signs of facial aging. | From baseline to 6-months post-Sculptra therapy

SECONDARY OUTCOMES:
Document the types and incidence of device adverse events with Sculptra Therapy (Injectable PLLA) | From baseline to 6-months post-Sculptra therapy

CONTACTS AND LOCATIONS:
Overall Officials: Mary Tzortzis, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Québec, Canada